CLINICAL TRIAL: NCT00100516
Title: Infrared Image Guided Minimally Invasive Live Donor Kidney Donation for Kidney Transplantation
Brief Title: Donor Recipient Kidney Function Following Open Surgical vs. Laparoscopic Kidney Donation
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050043; 05-DK-0043
Record Dates: First submitted 2004-12-31; First posted 2005-01-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Kidney Transplantation
Keywords: Renal; Allografts; Nephrectomy; Pneumoperitoneum; LaparoscopIC; Kidney Donation
MeSH Terms: conditions — Pneumoperitoneum

SUMMARY:
This study will evaluate the differences between open surgical kidney donation and laparoscopic kidney donation on kidney donors and recipients. Both procedures are standard surgeries used to remove kidneys for donation, and they are done equally often. Open surgical kidney donation involves removing the donor kidney through a 3- to 5-inch surgical incision. Laparoscopic donation involves making several small holes in the skin and removing the kidney through a larger hole, while directly watching the kidney with a camera. The study will correlate the effects of both procedures with donor and recipient kidney function, urine output, post-operative pain, and return to work after surgery.

Adults without kidney disease who are willing to donate a kidney to a patient enrolled in a clinical transplant protocol at the NIH Clinical Center may be eligible for this study. Donors and recipients must be enrolled in the NIDDK protocol, Live Donor Renal Donation for Allotransplantation (protocol #99-DK-0107).

Donors and patients undergo the following procedures:

* Infrared imaging (measurement of small differences in temperature using a special camera) during surgery to look at blood flow to the kidney during the operation (both donor and recipient surgical procedures). The pictures provide images of the blood vessels in the kidney and measure how the blood flow changes.
* Kidney biopsy (removal of a small piece of kidney tissue). The patient's failed kidney is biopsied once during transplant surgery when it is removed. The donor's kidney is biopsied twice - once during surgery to remove the organ from the donor and again after transplant into the recipient.
* Evaluations after surgery of post-operative urine output, blood pressure, and pain, and length of hospital stay and return to work.

DETAILED DESCRIPTION:
Laparoscopic techniques are increasingly being used for live donor nephrectomy for kidney transplantation. The technical methods have been rapidly adopted by the transplant community, but remain limited by the requirement for pneumoperitoneum, a technique that increases intra-abdominal pressure to gain surgical exposure. Pneumoperitoneum reduces renal cortical blood flow, potentially inducing ischemia associated factors that promote allograft rejection or attenuate post transplant renal function.

The aim of this study is to determine the effects of pneumoperitoneum used for minimally invasive donor nephrectomy on renal perfusion using infrared imaging. Our goals are to:

1. Analyze the effect of varying levels of pneumoperitoneum intraoperatively using infrared imaging;
2. Correlate the effects of both open and laparoscopic living donation with respect to transcriptional events, donor and recipient renal function, urine output, post-operative pain and return to work postoperatively;
3. Determine optimal conditions for procurement of renal allografts for subjects undergoing renal transplantation.

In this study, patients will be those who have been consented to kidney donation on the Live Donor Renal Donation for Allotransplantation (99-DK-0107). This study will represent the first such use of infrared imaging and the first prospective evaluation of strategies for living kidney donation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients enrolled in the Live Donor Renal Donation for Allotransplantation 99-DK-0107.

EXCLUSION CRITERIA:

Patients ineligible for this protocol will be excluded.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12-23; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Tarantino A. Why should we implement living donation in renal transplantation? Clin Nephrol. 2000 Apr;53(4):suppl 55-63. PMID 10809438